CLINICAL TRIAL: NCT01436812
Title: International Reveiw Board of Gachon Univerity Gil Hospital
Brief Title: Effect of Positive End Expiratory Pressure (PEEP) on Cerebral Oxymetry During Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Assistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GIRBA2551; GIRBA2551 (Registry Identifier: IRB of Gachon University Gil Hospital)
Record Dates: First submitted 2011-09-15; First posted 2011-09-20 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Cerebral Ischemia
Keywords: cerebral oxymetry; laparoscopy; PEEP
MeSH Terms: conditions — Brain Ischemia | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zero end-expiratory pressure (Placebo Comparator): not applying PEEP during operation just applying TV=IBW*6-8ml IBW = (male; 50+0.91[(Ht-cm)-152.4], female; 45.5 +0.91[(Ht-cm)-152.4], RR 8-12/min,
  Interventions: Procedure: positive end expiratory pressure
- positive end expiratory pressure (Active Comparator): applying PEEP 10cmH2O during operation just applying TV=IBW*6-8ml IBW = (male; 50+0.91[(Ht-cm)-152.4], female; 45.5 +0.91[(Ht-cm)-152.4], RR 8-12/min,
  Interventions: Procedure: zero end-expiratory pressure

INTERVENTIONS:
Procedure: zero end-expiratory pressure — positive end expiratory pressure 0 cm H2O during peumoperitoneum
  Other Names: ZEEP
  Arms: positive end expiratory pressure
Procedure: positive end expiratory pressure — PEEP 0 cmH2O
  Other Names: ZEEP
  Arms: zero end-expiratory pressure

SUMMARY:
The investigators hypothesized that positive end expiratory pressure (PEEP) would increase the regional oxygen saturation (rSO2).

DETAILED DESCRIPTION:
The investigators hypothesized that PEEP would increase the rSO2 during laparoscopic surgery by improving oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS I or II adult patient undergoing laparoscopic low anterior resection with Trendelenburg position

Exclusion Criteria:

* Patients with history of cerebrovascular disease, coronary occlusive disease and/or obesity (body mass index > 30) were excluded from this study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
cerebral ischemia | change from baseline in rSO2 at every events
  induction 10 min, Pneumoperitoneum 20 min, after PEEP apply 40 min, time of operation ending cerebral oxymetry, cerebral perfusion pressure record

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jeong Kwak, MD.PhD, Study Chair — Gachon University Gil Medical Center; Youn Yi Jo, MD.PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Hospital, Incheon, South Korea